CLINICAL TRIAL: NCT01875549
Title: Comparison Between Unilateral Versus Bilateral Stenting for Malignant Hilar Biliary Obstruction to Use a Large Cell Niti-S (LCD) Stent
Brief Title: Comparison Between Unilateral Versus Bilateral Stenting for Malignant Hilar Biliary Obstruction to Use a LCD Stent
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: Kwang Hyuck Lee (Other)
Responsible Party: Sponsor-Investigator, Kwang Hyuck Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-03-014-002
Record Dates: First submitted 2013-06-04; First posted 2013-06-12 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Obstruction of Biliary Tree; Cholangiocarcinoma; Hepatocellular Carcinoma; Malignant Lymphadenopathy; Gall Bladder Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular; Gallbladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unilateral stent insertion group (Active Comparator): the use of unilateral stent insertion in malignant hilar obstruction for using endoscopic retrograde cholangiopancreatography(ERCP)
  Interventions: Device: stent insertion; Procedure: Endoscopic retrograde cholangiopancreatoscopy(ERCP)
- Bilateral stent insertion group (Active Comparator): the use of bilateral stent insertion in malignant hilar obstruction for using endoscopic retrograde cholangiopancreatography(ERCP)
  Interventions: Device: stent insertion; Procedure: Endoscopic retrograde cholangiopancreatoscopy(ERCP)

INTERVENTIONS:
Device: stent insertion — to use a LCD stent at an unilateral or bilateral stent insertion
  Other Names: Niti-S large cell D-type biliary stent [LCD]
Procedure: Endoscopic retrograde cholangiopancreatoscopy(ERCP) — to use ERCP for a stent insertion in an obstructive biliary tract

SUMMARY:
Internal biliary drainage is an useful method for a control of jaundice and cholangitis to patients who had a malignant hilar obstruction due to hepatocellular carcinoma, cholangiocarcinoma, gall bladder cancer or metastatic lymphadenopathy.

Bilateral biliary drainage is more physiologic but technically difficult to compared with unilateral biliary drainage specially related to conformability and flexibility between using stents.

There are no prospective clinical trials compared with these internal biliary drainage methods in hilar malignant obstruction using metal stent.

Therefore, the investigators want to compare the clinical outcome of two method: Unilateral biliary stent and Bilateral biliary stent

ELIGIBILITY:
Inclusion Criteria:

* Age> 18
* diagnosis of malignancy in pathology or cytology
* jaundice(Total bilirubin)> 2.0 mg/dL
* Diagnosed malignant hilar invasion to CT or other image finding

Exclusion Criteria:

* bleeding tendency(INR>1.5)
* Pregnancy
* severe liver,kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Stent patency | up to 1year
  Participants will followed for the new obstruction(new jaundice) will occur.

SECONDARY OUTCOMES:
survival period | up to 1year
  Participants will followed for 1year.

OTHER OUTCOMES:
complication | up to 1year
  Participants will followed after stent insertion and observe a complication rate between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang hyuck Lee, PhD, Study Director — Division of Gastroenterology,Department of internal medicaion,samsung medical center,Sungkyunkwan University School of Medicine